CLINICAL TRIAL: NCT00593008
Title: A Phase 1 Study of Temsirolimus in Combination With Gemcitabine in Previously Untreated Metastatic Pancreatic Cancer
Brief Title: Temsirolimus in Combination With Gemcitabine in Previously Untreated Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Eunice L. Kwak, MD, PhD, Assistant in Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-115
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — temsirolimus; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Temsirolimus — Given intravenously every week of each 28-day cycle (days 1, 8, 15 and 22). Participants may continue to receive study treatment as long as their tumor is responding and they don't experience any serious side effects.
Drug: Gemcitabine — Given intravenously every other week of each 28-day cycle.

SUMMARY:
The purpose of this research study is to try to define the highest doses of temsirolimus and gemcitabine that can be used safely in combination to treat advanced pancreatic cancer. Gemcitabine is a standard chemotherapy used for the treatment of pancreatic cancer.

DETAILED DESCRIPTION:
* Because this is a study to determine the highest doses of temsirolimus and gemcitabine that can be given safely together, groups of 3 subjects will be treated at gradually increasing doses of the drugs. Each group of 3 subjects must complete 4 weeks of treatment (1 cycle) before the following group of 3 subjects can start treatment at the higher dose of drug.
* Temsirolimus will be given intravenously every week of the 28 day treatment cycle (days 1, 8, 15, 22). Gemcitabine will be given intravenously every other week of the treatment cycle (days 1. 15).
* During the study, participants will have weekly clinic visits where the following tests and procedures may be performed: Physical exam; vital signs; urine test; blood tests.
* A CT scan will be performed after every 2 cycles (8 weeks) to assess teh response of the tumor to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated metastatic pancreatic adenocarcinoma, histologically proven.
* Measurable disease by RECIST criteria
* ECOG Performance Status 0 or 1
* Male or female, 18 years of age or older
* Life expectancy of >/= 12 weeks
* AST and ALT </= 2.5 x ULN
* Total bilirubin </= 1.5 x ULN
* Serum albumin >/= 2.5g/dL
* Absolute neutrophil count >/= 1500/mm3; platelets >/= 100,000/mm3; hemoglobin >/= 9.0 g/dL
* Serum creatinine </= 1.5 x ULN
* Subjects with diabetes must have adequate glycemic control, with fasting serum glucose </= 1.5 x ULN
* Female patients of childbearing age and male patients with partners of childbearing age must agree to use adequate birth control measures during the course of the study and for at least one month following withdrawal from the study

Exclusion Criteria:

* Previously treatment with gemcitabine or chemoradiation
* Diagnosis of a second malignancy within the last 3 years, except for adequately treated basal cell carcinoma or squamous cell skin cancer
* Ongoing cardiac dysrhythmias of NCI CTCAE grade >/= 2, atrial fibrillation, QTc prolongation to > 450 msec for males and >470 msec for females
* Known immunodeficiency disorders or active infections requiring treatment
* Pregnancy or breastfeeding
* Known brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease
* Prior radiation therapy or major surgery within 4 weeks of study entry
* Prior radiation therapy to > 25% of the bone marrow
* Subjects receiving other experimental or alternative therapies during the course of the trial will be excluded
* History of prior hypersensitivity to polysorbate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicities and maximal tolerated doses of gemcitabine combined with temsirolimus | 2 years
To determine whether order of administration of the drugs affects the above | 2 years
To determine the dosing regimen appropriate for Phase 2 studies of the combination | 2 years

SECONDARY OUTCOMES:
To document objective response rate and progression-free survival in patients treated with this combination

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Kwak, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States